CLINICAL TRIAL: NCT04229225
Title: A Double-Blind, Randomized, Placebo-Controlled Study of Single and Repeat Dose Administration of UBX0101 in Moderate to Severe, Painful Osteoarthritis of the Knee
Brief Title: A Study of Single and Repeat Dose Administration of UBX0101 in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unity Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UBX0101-MUS-102
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-04

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Painful Osteoarthritis; Osteoarthritis, Knee; Senescence
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UBX0101 single dose (SD) (Experimental): Cohort 1 (n=18): UBX0101 8.0 mg or placebo IA at Week 0
  Patients will be randomized in a 2:1 ratio to UBX0101 and placebo
  Interventions: Drug: UBX0101; Other: Placebo
- UBX0101 repeat dose (RD) (Experimental): Cohort 2 (n=18): UBX0101 4.0 mg or placebo IA at Weeks 0 and 4
  Patients will be randomized in a 2:1 ratio to UBX0101 and placebo
  Interventions: Drug: UBX0101; Other: Placebo

INTERVENTIONS:
Drug: UBX0101 — Investigational drug intra-articular (IA) injection
Other: Placebo — Placebo intra-articular (IA) injection

SUMMARY:
A study to assess safety, tolerability and clinical effects of single and repeat dose intra-articular administration of UBX0101 in patients with moderate to severe painful knee osteoarthritis (OA).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted as two parallel cohorts to assess the safety, tolerability, and clinical effects of single dose (SD) and repeat dose (RD) intra-articular (IA) administration of UBX0101 in patients with symptomatic knee osteoarthritis (OA).

Approximately 36 patients will be randomly assigned to either Cohort 1 (SD) or Cohort 2 (RD) (18 patients per treatment cohort) and further randomized in a 2:1 ratio to UBX0101 and placebo in each cohort.

The primary objective of the study is to evaluate the safety and tolerability of SD and RD IA administration of UBX0101 over 24 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients who are ambulatory with a diagnosis of OA of the knee and who have moderate to severe knee pain as measured on the 11-point (0-10) average daily pain NRS.
* Kellgren-Lawrence grade of 1-4 on a weight-bearing radiograph of target knee.
* Patients aged ≥ 40 and ≤ 85 years.
* Patients are permitted but not required to use an oral NSAID, serotonin, and norepinephrine reuptake inhibitors (SNRIs), tramadol, or acetaminophen, provided that they have been taking a stable dose and regimen of medication for at least 4 weeks prior to Screening.

Key Exclusion Criteria:

* Patients with any condition, including laboratory or imaging findings and findings in the medical history or in the pre-study assessments, that in the opinion of the Investigator or the Medical Monitor constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation or prevent the patient from fully participating in all aspects of the study.
* Patients with a body mass index (BMI) ≥40 kg/m².
* Patients with fibromyalgia.
* Systemic autoimmune disease with musculoskeletal involvement or any history of a systemic inflammatory arthritis.
* Patients who have received IA treatment in the target knee with steroids or hyaluronic acid derivatives within the last 16 weeks prior to Screening, or with extended-release corticosteroid (e.g., Zilretta®) within the last 20 weeks.
* Patients who are using a topical NSAID or topical analgesics on the target knee.
* Patients who have used opioid analgesics (other than tramadol), marijuana or marijuana-derived products (e.g., cannabidiol), and topical capsaicin on the target knee within 8 weeks prior to Screening.
* Patients with a history of traumatic knee injury to the target knee, including, but not limited to, patients with meniscal root tear, within 2 years of study entry.
* Patients who have undergone diagnostic arthroscopy to the target knee in the previous 6 months.
* Patients who have undergone arthroscopic surgery (including microfracture and meniscectomy) on the target knee in the last 2 years prior to the Screening visit or are anticipated to have arthroscopic surgery on either knee at any time during the study period.
* Patients with a history of previous total or partial knee arthroplasty in the target knee.
* Patients with an effusion at the Screening visit, which, in the opinion of the Investigator following examination and discussions with the patient, requires drainage for symptom relief.
* Patients who have had regenerative joint procedures on any joint, including, but not limited to, platelet-rich plasma injections, stem cell transplantation, autologous chondrocyte transplantation, or mosaicplasty.
* Patients with secondary arthritis that involves the target knee or would confound assessments of knee OA.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a single and repeat dose intra-articular administration of UBX0101 evaluated by the incidence of serious and non-serious adverse events | Baseline to Week 24

SECONDARY OUTCOMES:
Plasma UBX0101 drug concentrations following IA administration | 1, 2, and 4 hours post-dose for both cohorts on Day 1 and at 1, 2, and 4 hours post-dose at Week 4 for Cohort 2 only
Change from baseline to Week 12 of the Western Ontario and McMaster Universities Osteoarthritis Index pain subscale (WOMAC-A) score in patients receiving UBX0101 versus those receiving placebo | Baseline to Week 12
  WOMAC-A is assessed by a Likert scale on a range from 0 (none) to 4 (extreme), with higher scores indicating higher levels of pain
Change from baseline to Week 24 of the WOMAC-A score over time in patients receiving UBX0101 versus those receiving placebo | Baseline to Week 24
  WOMAC-A is assessed by a Likert scale on a range from 0 (none) to 4 (extreme), with higher scores indicating higher levels of pain
Change from baseline to Week 12 of the Western Ontario and McMaster Universities Osteoarthritis Index function subscale (WOMAC-C) score in patients receiving UBX0101 versus those receiving placebo | Baseline to Week 12
  WOMAC-C is assessed by a Likert scale on a range from 0 (none) to 4 (extreme), with higher scores indicating higher levels of physical disability
Change from baseline to Week 12 of the weekly mean of the average daily pain (ADP) intensity scores on the 11-point numeric rating scale (NRS) in patients receiving UBX0101 versus those receiving placebo | Baseline to Week 12
  ADP is assessed by NRS on a range from 0 (no pain) to 10 (worst pain imaginable), with higher scores indicating higher levels of pain

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Unity Biotechnology
Locations (7):
- United States (7):
  - Premier Medical Associates, The Villages, Florida
  - Drug Studies America, Marietta, Georgia
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - Rochester Clinical Research, Inc., Rochester, New York
  - Arcis Healthcare LLC dba Lowcountry Orthopaedics and Sports Medicine, North Charleston, South Carolina
  - First Surgical Hospital, Bellaire, Texas